CLINICAL TRIAL: NCT00215657
Title: An Open-Label, Multi-Center, Extension Study Investigating the Long-Term Safety and Tolerability of Repeat Doses of FE200486 in Prostate Cancer Patients
Brief Title: Extension Study Investigating the Long-Term Safety and Tolerability of Repeat Doses of FE200486 in Prostate Cancer Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The doses were not effective in maintaining testosterone suppression
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FE200486 CS07A
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Results first posted 2009-06-12 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2011-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Degarelix 120 mg (20 mg/mL) (Experimental): Degarelix 120 mg (20 mg/mL)
  Interventions: Drug: Degarelix
- Degarelix 120 mg (40 mg/mL) (Experimental): Degarelix 120 mg (40 mg/mL)
  Interventions: Drug: Degarelix
- Degarelix 160 mg (40 mg/mL) (Experimental): Degarelix 160 mg (40 mg/mL)
  Interventions: Drug: Degarelix
- Degarelix 200 mg (40 mg/mL) (Experimental): Degarelix 200 mg (40 mg/mL)
  Interventions: Drug: Degarelix
- Degarelix 200 mg (60 mg/mL) (Experimental): Degarelix 200 mg (60 mg/mL)
  Interventions: Drug: Degarelix
- Degarelix 240 mg (40 mg/mL) (Experimental): Degarelix 240 mg (40 mg/mL)
  Interventions: Drug: Degarelix
- Degarelix 240 mg (60 mg/mL) (Experimental): Degarelix 240 mg (60 mg/mL)
  Interventions: Drug: Degarelix
- Degarelix 320 mg (60 mg/mL) (Experimental): Degarelix 320 mg (60 mg/mL)
  Interventions: Drug: Degarelix

INTERVENTIONS:
Drug: Degarelix — Degarelix 120 mg (20 mg/mL). Participants received same dose as in main study (FE200486 CS07; NCT00818623). Administration intervals were individualised for each participant (based on the duration of testosterone suppression in study FE200486 CS07).
  Other Names: FE200486
  Arms: Degarelix 120 mg (20 mg/mL)
Drug: Degarelix — Degarelix 120 mg (40 mg/mL). Participants received same dose as in main study (FE200486 CS07; NCT00818623). Administration intervals were individualised for each participant (based on the duration of testosterone suppression in study FE200486 CS07).
  Other Names: FE200486
  Arms: Degarelix 120 mg (40 mg/mL)
Drug: Degarelix — Degarelix 160 mg (40 mg/mL). Participants received same dose as in main study (FE200486 CS07; NCT00818623). Administration intervals were individualised for each participant (based on the duration of testosterone suppression in study FE200486 CS07).
  Other Names: FE200486
  Arms: Degarelix 160 mg (40 mg/mL)
Drug: Degarelix — Degarelix 200 mg (40 mg/mL). Participants received same dose as in main study (FE200486 CS07; NCT00818623). Administration intervals were individualised for each participant (based on the duration of testosterone suppression in study FE200486 CS07).
  Other Names: FE200486
  Arms: Degarelix 200 mg (40 mg/mL)
Drug: Degarelix — Degarelix 200 mg (60 mg/mL). Participants received same dose as in main study (FE200486 CS07; NCT00818623). Administration intervals were individualised for each participant (based on the duration of testosterone suppression in study FE200486 CS07).
  Other Names: FE200486
  Arms: Degarelix 200 mg (60 mg/mL)
Drug: Degarelix — Degarelix 240 mg (40 mg/mL). Participants received same dose as in main study (FE200486 CS07; NCT00818623). Administration intervals were individualised for each participant (based on the duration of testosterone suppression in study FE200486 CS07).
  Other Names: FE200486
  Arms: Degarelix 240 mg (40 mg/mL)
Drug: Degarelix — Degarelix 240 mg (60 mg/mL). Participants received same dose as in main study (FE200486 CS07; NCT00818623). Administration intervals were individualised for each participant (based on the duration of testosterone suppression in study FE200486 CS07).
  Other Names: FE200486
  Arms: Degarelix 240 mg (60 mg/mL)
Drug: Degarelix — Degarelix 320 mg (60 mg/mL). Participants received same dose as in main study (FE200486 CS07; NCT00818623). Administration intervals were individualised for each participant (based on the duration of testosterone suppression in study FE200486 CS07).
  Other Names: FE200486
  Arms: Degarelix 320 mg (60 mg/mL)

SUMMARY:
An Open-Label, Multi-Center, Extension Study Investigating the Long-Term Safety and Tolerability of Repeat Doses of FE200486 in Prostate Cancer Patients

DETAILED DESCRIPTION:
Degarelix was not FDA regulated at the time of the trial. After completion of the trial degarelix has been approved by the FDA and is thus an FDA regulated intervention (FDA regulated intervention is therefore ticked "YES").

The data include participants from both the main study (FE200486 CS07; NCT00818623) and the extension study FE200486 CS07A.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18 or over
* Histologically proven adenocarcinoma of the prostate (all stages) in whom endocrine treatment was indicated (except neoadjuvant hormonal therapy)
* Has completed Study FE200486 CS07
* Has not met a withdrawal criteria at Visit 9 (day 28) in Study FE200486 CS07

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2003-03; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who responded to degarelix in FE200486 CS07 (NCT00818623) were eligible to enroll into this extension study with the intention of continuing treatment until degarelix became commercially available or until the study was discontinued. Participants received the same dose of degarelix as they received in FE200486 CS07.
Pre-assignment Details: 180 participants started the main study CS07 and 172 participants received degarelix treatment (intention-to-treat population). Of these, 131 participants were recruited into the extension study CS07A
Groups:
- Degarelix 120mg (20mg/mL): Degarelix 120 mg (20 mg/mL)
- Degarelix 120mg (40mg/mL): Degarelix 120 mg (40 mg/mL)
- Degarelix 160mg (40mg/mL): Degarelix 160 mg (40 mg/mL)
- Degarelix 200mg (40mg/mL): Degarelix 200 mg (40 mg/mL)
- Degarelix 200mg (60mg/mL): Degarelix 200 mg (60 mg/mL)
- Degarelix 240mg (40mg/mL): Degarelix 240 mg (40 mg/mL)
- Degarelix 240mg (60mg/mL): Degarelix 240 mg (60 mg/mL)
- Degarelix 320mg (60mg/mL): Degarelix 320 mg (60 mg/mL)
Period: Overall Study
Arm/Group | Degarelix 120mg (20mg/mL) | Degarelix 120mg (40mg/mL) | Degarelix 160mg (40mg/mL) | Degarelix 200mg (40mg/mL) | Degarelix 200mg (60mg/mL) | Degarelix 240mg (40mg/mL) | Degarelix 240mg (60mg/mL) | Degarelix 320mg (60mg/mL)
Started | 26 | 12 | 13 | 24 | 27 | 24 | 27 | 27
Intention-to-treat Population | 25 | 12 | 12 | 24 | 24 | 24 | 24 | 27
Started FE200486 CS07A | 20 | 6 | 7 | 24 | 17 | 20 | 14 | 23
Completed | 4 (Participants ongoing at the time of study closure were considered to have completed the study.) | 1 | 2 | 6 | 4 | 4 | 4 | 11
Not Completed | 22 | 11 | 11 | 18 | 23 | 20 | 23 | 16
Not completed — Adverse Event | 5 | 1 | 3 | 0 | 3 | 1 | 0 | 3
Not completed — Withdrawal by Subject | 6 | 3 | 3 | 1 | 6 | 1 | 10 | 3
Not completed — Insuff prostate specific antigen resp | 3 | 2 | 2 | 2 | 1 | 2 | 3 | 2
Not completed — Insufficient testosterone response | 5 | 4 | 1 | 12 | 8 | 12 | 4 | 7
Not completed — Other | 3 | 1 | 2 | 3 | 5 | 4 | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Degarelix 120mg (20mg/mL) | Degarelix 120mg (40mg/mL) | Degarelix 160mg (40mg/mL) | Degarelix 200mg (40mg/mL) | Degarelix 200mg (60mg/mL) | Degarelix 240mg (40mg/mL) | Degarelix 240mg (60mg/mL) | Degarelix 320mg (60mg/mL) | Total
Number analyzed (Participants) | 25 | 12 | 12 | 24 | 24 | 24 | 24 | 27 | 172
Age, Categorical [Count of Participants; unit: Participants] — Intention-to-treat (ITT) population.
  Participants
    <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 7 | 0 | 2 | 2 | 4 | 2 | 6 | 6 | 29
    >=65 years | 18 | 12 | 10 | 22 | 20 | 22 | 18 | 21 | 143
Age Continuous [Mean (Standard Deviation); unit: years] — ITT population.
  years | 70.0 (10.3) | 73.8 (3.97) | 70.1 (8.08) | 74.3 (6.48) | 71.5 (8.27) | 73.1 (5.96) | 71.7 (9.54) | 71.1 (6.87) | 71.9 (7.83)
Sex: Female, Male [Count of Participants; unit: Participants] — ITT population.
  Participants
    Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Male | 25 | 12 | 12 | 24 | 24 | 24 | 24 | 27 | 172
Race/Ethnicity, Customized [Number; unit: participants] — ITT population.
  participants
    Caucasian | 25 | 12 | 12 | 24 | 24 | 24 | 24 | 27 | 172
Curative intent [Number; unit: participants] — ITT population. A curative intent of Yes refers to participants who have been castrated via radical prostatectomy or radiotherapy.
  participants
    Yes | 0 | 0 | 2 | 3 | 1 | 0 | 0 | 1 | 7
    No | 25 | 12 | 10 | 21 | 23 | 24 | 24 | 26 | 165
Gleason score [Number; unit: participants] — ITT population. The Gleason score is a system of grading the aggressiveness of the prostate cancer and how fast it is likely to grow and spread. Scale is 2-10, with low numbers being the least aggressive and 10 being the most aggressive.
  participants
    2-4 | 4 | 0 | 2 | 1 | 5 | 2 | 5 | 12 | 31
    5-6 | 4 | 7 | 5 | 6 | 3 | 6 | 6 | 6 | 43
    7-10 | 17 | 5 | 5 | 17 | 16 | 16 | 13 | 9 | 98
Stage of prostate cancer [Number; unit: participants] — ITT population. Prostate cancer stage was classified to describe the extent of cancer. Localized refers to tumors without involvement of lymph nodes or metastasis. Advanced localized can be larger tumors that may involve the lymph nodes but no metastasis. Metastatic are more advanced cancers that are spreading beyond the original tumor.
  participants
    Localized | 10 | 1 | 3 | 3 | 1 | 6 | 8 | 14 | 46
    Locally advanced | 6 | 6 | 5 | 14 | 8 | 10 | 5 | 9 | 63
    Metastatic | 9 | 3 | 4 | 6 | 12 | 6 | 10 | 2 | 52
    Not classifiable | 0 | 2 | 0 | 1 | 3 | 2 | 1 | 2 | 11
Body mass index [Mean (Standard Deviation); unit: kilogram per square meter] — ITT population.
  kilogram per square meter | 26.2 (2.97) | 26.6 (4.58) | 26.3 (3.74) | 25.9 (2.99) | 24.5 (2.92) | 26.9 (3.18) | 24.8 (2.72) | 27.1 (3.63) | 26.0 (3.32)
Time since prostate cancer diagnosis [Mean (Standard Deviation); unit: days] — ITT population.
  days | 83 (157) | 66 (53) | 222 (328) | 146 (298) | 252 (560) | 303 (837) | 121 (425) | 47 (54) | 156 (439)
Weight [Mean (Standard Deviation); unit: kilogram] — ITT population.
  kilogram | 77.8 (12.4) | 82.2 (12.1) | 80.7 (11.8) | 78.2 (13.7) | 74.2 (9.88) | 81.5 (10.7) | 73.5 (9.55) | 81.7 (11.1) | 78.4 (11.6)

OUTCOME MEASURES:

1. Primary Outcome: Liver Function Tests
Description: The figures present the number of participants who had abnormal (defined as above upper limit of normal range (ULN)) alanine aminotransferase (ALT) levels, aspartate aminotransferase levels, and bilirubin levels plus the number of participants who had ALT increases >3x ULN and ALT increases >3x ULN with concurrently increased bilirubin >1.5 ULN.
Time Frame: 3 years
Population: The data include patients from both the main study (FE200486 CS07) and the extension study FE200486 CS07A
Measure: Number; unit: participants
Arm/Group | Degarelix 120mg (20mg/mL) | Degarelix 120mg (40mg/mL) | Degarelix 160mg (40mg/mL) | Degarelix 200mg (40mg/mL) | Degarelix 200mg (60mg/mL) | Degarelix 240mg (40mg/mL) | Degarelix 240mg (60mg/mL) | Degarelix 320mg (60mg/mL)
Number analyzed (Participants) | 25 | 12 | 12 | 24 | 24 | 24 | 24 | 27
participants
  Abnormal alanine aminotransferase (ALAT) | 11 | 4 | 3 | 7 | 7 | 7 | 7 | 9
  Abnormal aspartate aminotransferase | 9 | 4 | 2 | 6 | 8 | 6 | 6 | 7
  Abnormal bilirubin | 4 | 2 | 0 | 2 | 0 | 2 | 0 | 1
  ALAT >3x ULN | 4 | 0 | 0 | 0 | 0 | 2 | 1 | 1
  ALAT >3x ULN, bilirubin >2x ULN | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0

2. Primary Outcome: Participants With Markedly Abnormal Change in Vital Signs and Body Weight
Description: Vital signs and body weight included incidence of markedly abnormal changes in blood pressure (systolic and diastolic), pulse, and body weight at the end of trial as compared to baseline. The table presents the number of patients in each group with normal baseline and markedly abnormal value post-baseline.
Time Frame: 3 years
Population: These data include patients from the main study (FE200486 CS07) and the extension study (FE200486 CS07A).
Measure: Number; unit: participants
Arm/Group | Degarelix 120mg (20mg/mL) | Degarelix 120mg (40mg/mL) | Degarelix 160mg (40mg/mL) | Degarelix 200mg (40mg/mL) | Degarelix 200mg (60mg/mL) | Degarelix 240mg (40mg/mL) | Degarelix 240mg (60mg/mL) | Degarelix 320mg (60mg/mL)
Number analyzed (Participants) | 25 | 12 | 12 | 24 | 24 | 24 | 24 | 27
participants
  Diastolic blood pressure <=50 and decrease >=15 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Diastolic blood pressure >=105 and increase >=15 | 2 | 0 | 1 | 1 | 2 | 1 | 1 | 2
  Systolic blood pressure <=90 and decrease >=20 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Systolic blood pressure >=180 and increase >=20 | 0 | 0 | 2 | 5 | 2 | 6 | 2 | 3
  Heart rate <=50 and decrease >=15 | 1 | 1 | 2 | 0 | 2 | 1 | 1 | 1
  Heart rate >=120 and increase >=15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Body weight decrease of >=7 percent | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 1
  Body weight increase of >=7 percent | 4 | 2 | 3 | 9 | 3 | 8 | 7 | 2

ADVERSE EVENTS:
Arm/Group | Degarelix 120mg (20mg/mL) | Degarelix 120mg (40mg/mL) | Degarelix 160mg (40mg/mL) | Degarelix 200mg (40mg/mL) | Degarelix 200mg (60mg/mL) | Degarelix 240mg (40mg/mL) | Degarelix 240mg (60mg/mL) | Degarelix 320mg (60mg/mL)
Serious Adverse Events (participants affected / at risk) | 8 | 4 | 3 | 7 | 8 | 5 | 3 | 9
Other Adverse Events (participants affected / at risk) | 18 | 10 | 9 | 24 | 17 | 22 | 12 | 19
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Degarelix 120mg (20mg/mL) | Degarelix 120mg (40mg/mL) | Degarelix 160mg (40mg/mL) | Degarelix 200mg (40mg/mL) | Degarelix 200mg (60mg/mL) | Degarelix 240mg (40mg/mL) | Degarelix 240mg (60mg/mL) | Degarelix 320mg (60mg/mL)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Cardiac failure (Cardiac disorders) | 1/25 (2) | 0/12 (0) | 0/12 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/27 (1)
Angina unstable (Cardiac disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Myocardial infarction (Cardiac disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/27 (1)
Myocardial ischemia (Cardiac disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/27 (1)
Vertigo (Ear and labyrinth disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Inguinal hernia (Gastrointestinal disorders) | 1/25 (1) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Gastritis (Gastrointestinal disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/27 (1)
Mallory-weiss syndrome (Gastrointestinal disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Mechanical ileus (Gastrointestinal disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Disease progression (General disorders) | 1/25 (1) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Pyrexia (General disorders) | 1/25 (1) | 0/12 (0) | 1/12 (1) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Asthenia (General disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/27 (1)
Chest pain (General disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Cholelithiasis (Hepatobiliary disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/27 (0)
Sepsis (Infections and infestations) | 1/25 (1) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Urinary tract infection (Infections and infestations) | 1/25 (1) | 0/12 (0) | 0/12 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Bronchitis (Infections and infestations) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Erysipelas (Infections and infestations) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Infection (Infections and infestations) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Neutropenic sepsis (Infections and infestations) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/27 (1)
Pneumonia (Infections and infestations) | 1/25 (1) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/27 (0)
Caustic injury (Injury, poisoning and procedural complications) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/27 (1)
Contusion (Injury, poisoning and procedural complications) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/27 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Gamma-glutamyltransferase increased (Investigations) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/27 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1/25 (1) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1/25 (1) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/25 (1) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Bladder transitional cell carcinoma stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/25 (1) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/27 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/25 (2) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 1/24 (1) | 0/27 (0)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Cerebral infarction (Nervous system disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Epilepsy (Nervous system disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Parkinson's disease (Nervous system disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Spinal cord compression (Nervous system disorders) | 1/25 (1) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Completed suicide (Psychiatric disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Renal failure acute (Renal and urinary disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 2/24 (2) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Urinary retention (Renal and urinary disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Haematuria (Renal and urinary disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 1/24 (1) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/27 (0)
Hydronephrosis (Renal and urinary disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1/25 (1) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1/25 (1) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Thrombosis (Vascular disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Acute myocardial infarction (Cardiac disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/27 (0)
Vomiting (Gastrointestinal disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/27 (0)
Condition aggravated (General disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Oedema (General disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Hepatitis toxic (Hepatobiliary disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/27 (1)
Gangrene (Infections and infestations) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/27 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1/25 (1) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/27 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Areflexia (Nervous system disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Ischaemic stroke (Nervous system disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/27 (1)
Paraplegia (Nervous system disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/27 (0)
Depression (Psychiatric disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/27 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1/25 (1) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Amputation revision (Surgical and medical procedures) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Deep vein thrombosis (Vascular disorders) | 1/25 (1) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Hypertension (Vascular disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/27 (0)
Angina pectoris (Cardiac disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/27 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Degarelix 120mg (20mg/mL) | Degarelix 120mg (40mg/mL) | Degarelix 160mg (40mg/mL) | Degarelix 200mg (40mg/mL) | Degarelix 200mg (60mg/mL) | Degarelix 240mg (40mg/mL) | Degarelix 240mg (60mg/mL) | Degarelix 320mg (60mg/mL)
Anaemia (Blood and lymphatic system disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 2/24 (2) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/27 (0)
Angina pectoris (Cardiac disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 1/24 (1) | 1/24 (1) | 1/24 (1) | 2/27 (2)
Arrhytmia (Cardiac disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Atrial fibrillation (Cardiac disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/27 (0)
Phimosis (Congenital, familial and genetic disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Cataract (Eye disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 2/24 (2) | 1/27 (1)
Glaucoma (Eye disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/27 (0)
Constipation (Gastrointestinal disorders) | 2/25 (2) | 0/12 (0) | 0/12 (0) | 1/24 (1) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 1/27 (1)
Nausea (Gastrointestinal disorders) | 0/25 (0) | 2/12 (2) | 1/12 (1) | 3/24 (4) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/27 (0)
Abdominal pain (Gastrointestinal disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 1/24 (1) | 0/27 (0)
Diarrhoea (Gastrointestinal disorders) | 1/25 (1) | 1/12 (1) | 0/12 (0) | 4/24 (4) | 0/24 (0) | 1/24 (1) | 1/24 (1) | 1/27 (1)
Vomiting (Gastrointestinal disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 1/24 (2) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/27 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 2/24 (2) | 0/24 (0) | 0/27 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Dyspepsia (Gastrointestinal disorders) | 1/25 (1) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/27 (0)
Gastritis (Gastrointestinal disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Pyrexia (General disorders) | 2/25 (2) | 0/12 (0) | 1/12 (2) | 2/24 (3) | 0/24 (0) | 2/24 (4) | 1/24 (2) | 1/27 (1)
Fatigue (General disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 5/24 (7) | 2/24 (2) | 0/24 (0) | 0/24 (0) | 1/27 (1)
Injection site erythema (General disorders) | 0/25 (0) | 1/12 (1) | 1/12 (2) | 4/24 (4) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/27 (1)
Injection site induration (General disorders) | 1/25 (1) | 0/12 (0) | 1/12 (1) | 2/24 (2) | 0/24 (0) | 1/24 (2) | 0/24 (0) | 0/27 (0)
Injection site swelling (General disorders) | 1/25 (1) | 0/12 (0) | 1/12 (2) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Injection site pain (General disorders) | 1/25 (1) | 2/12 (2) | 1/12 (1) | 2/24 (2) | 2/24 (2) | 2/24 (2) | 0/24 (0) | 0/27 (0)
Oedema peripheral (General disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 1/24 (1) | 2/24 (3) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Chills (General disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 2/24 (2) | 0/24 (0) | 0/27 (0)
Feeling of body temperature change (General disorders) | 2/25 (3) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Injection site pruritus (General disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 2/24 (2) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Injection site reaction (General disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Urinary tract infection (Infections and infestations) | 3/25 (4) | 0/12 (0) | 1/12 (1) | 4/24 (6) | 2/24 (2) | 4/24 (5) | 4/24 (5) | 2/27 (2)
Nasopharyngitis (Infections and infestations) | 1/25 (1) | 3/12 (3) | 0/12 (0) | 4/24 (4) | 0/24 (0) | 2/24 (2) | 0/24 (0) | 1/27 (1)
Influenza (Infections and infestations) | 1/25 (1) | 1/12 (1) | 0/12 (0) | 1/24 (2) | 0/24 (0) | 1/24 (1) | 1/24 (1) | 0/27 (0)
Injection site abscess (Infections and infestations) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 2/27 (2)
Localised infection (Infections and infestations) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Nail infection (Infections and infestations) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Oral fungal infection (Infections and infestations) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Sinusitis (Infections and infestations) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Injury (Injury, poisoning and procedural complications) | 0/25 (0) | 1/12 (4) | 1/12 (1) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Blood alkaline phosphatase increased (Investigations) | 4/25 (5) | 1/12 (2) | 0/12 (0) | 2/24 (3) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 1/27 (1)
Alanine aminotranseferases increased (Investigations) | 4/25 (5) | 1/12 (3) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/27 (1)
Gamma-glutamyltransferase increased (Investigations) | 3/25 (4) | 1/12 (3) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 1/24 (3) | 0/24 (0) | 1/27 (1)
Weight decreased (Investigations) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 1/24 (1) | 2/24 (2) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Aspartate aminotransferase increased (Investigations) | 3/25 (3) | 1/12 (3) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Blood creatinine increased (Investigations) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 2/24 (2) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/27 (0)
Hepatic enzyme increased (Investigations) | 1/25 (1) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 2/24 (2) | 0/24 (0) | 0/27 (0)
White blood cells urine positive (Investigations) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Blood pressure increased (Investigations) | 1/25 (1) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 2/27 (3)
Lymphocyte count decreased (Investigations) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Prostatic specific antigen increased (Investigations) | 1/25 (1) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1/25 (1) | 1/12 (2) | 0/12 (0) | 5/24 (5) | 3/24 (4) | 3/24 (5) | 2/24 (2) | 1/27 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2/25 (2) | 0/12 (0) | 2/12 (2) | 2/24 (2) | 2/24 (2) | 1/24 (4) | 1/24 (1) | 2/27 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1/25 (1) | 0/12 (0) | 0/12 (0) | 1/24 (2) | 3/24 (3) | 1/24 (1) | 1/24 (1) | 1/27 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1/25 (1) | 0/12 (0) | 0/12 (0) | 2/24 (2) | 0/24 (0) | 1/24 (1) | 1/24 (1) | 0/27 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 2/25 (3) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 1/24 (1) | 0/27 (0)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/25 (2) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/27 (0)
Dizziness (Nervous system disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 3/24 (3) | 0/24 (0) | 0/24 (0) | 3/24 (3) | 0/27 (0)
Headache (Nervous system disorders) | 1/25 (1) | 2/12 (2) | 0/12 (0) | 4/24 (6) | 0/24 (0) | 3/24 (3) | 0/24 (0) | 0/27 (0)
Anosmia (Nervous system disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Insomnia (Psychiatric disorders) | 3/25 (3) | 0/12 (0) | 1/12 (1) | 4/24 (4) | 1/24 (1) | 0/24 (0) | 1/24 (2) | 0/27 (0)
Haematuria (Renal and urinary disorders) | 0/25 (0) | 0/12 (0) | 2/12 (3) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Pollakiuria (Renal and urinary disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 1/24 (2) | 1/24 (1) | 2/24 (2) | 1/24 (1) | 0/27 (0)
Cystitis noninfective (Renal and urinary disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Nocturia (Renal and urinary disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 3/24 (3) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2/25 (2) | 2/12 (2) | 0/12 (0) | 1/24 (1) | 2/24 (2) | 0/24 (0) | 2/24 (2) | 0/27 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2/25 (2) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6/25 (6) | 2/12 (2) | 1/12 (1) | 5/24 (6) | 5/24 (5) | 5/24 (5) | 2/24 (2) | 3/27 (3)
Erythema (Skin and subcutaneous tissue disorders) | 0/25 (0) | 0/12 (0) | 1/12 (2) | 1/24 (2) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/27 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/27 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/24 (2) | 0/27 (0)
Hot flush (Vascular disorders) | 4/25 (4) | 1/12 (1) | 3/12 (4) | 12/24 (14) | 6/24 (6) | 9/24 (9) | 4/24 (5) | 12/27 (13)
Hypertension (Vascular disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 2/24 (2) | 1/24 (1) | 0/27 (0)
Bradycardia (Cardiac disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Vertigo (Ear and labyrinth disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 2/24 (2) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/27 (0)
Haemorrhoids (Gastrointestinal disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 2/24 (2) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Inguinal hernia (Gastrointestinal disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Anal fissure (Gastrointestinal disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Stomach discomfort (Gastrointestinal disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Chest pain (General disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 2/24 (2) | 0/24 (0) | 0/27 (0)
Cystitis (Infections and infestations) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 1/27 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/27 (0)
Nervousness (Psychiatric disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Nightmare (Psychiatric disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/27 (0)
Prostatitis (Reproductive system and breast disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/27 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1/25 (1) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0/25 (0) | 1/12 (2) | 0/12 (0) | 1/24 (1) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Flushing (Vascular disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Hypoaesthesia (Nervous system disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript.